CLINICAL TRIAL: NCT06533865
Title: Romosozumab as an Adjunct to Physiologic Estrogen Replacement in Adolescents and Young Adults With Functional Hypothalamic Amenorrhea
Brief Title: Romosozumab as an Adjunct to Physiologic Estrogen Replacement in Functional Hypothalamic Amenorrhea
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024P000273
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-03

CONDITIONS: FHA (Functional Hypothalamic Amenorrhea)
MeSH Terms: interventions — romosozumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Romosozumab (Experimental): Participants with functional hypothalamic amenorrhea randomized to romosozumab.
  Interventions: Drug: Romosozumab; Drug: Zoledronic acid
- Placebo (Placebo Comparator): Participants with functional hypothalamic amenorrhea randomized to placebo.
  Interventions: Drug: Placebo; Drug: Zoledronic acid
- Healthy Controls (No Intervention): Healthy controls (girls and women with regular menstrual periods)

INTERVENTIONS:
Drug: Romosozumab — Six monthly subcutaneous injections. This group will also receive a 100-microgram transdermal estradiol patch applied twice weekly, and 200 mg of oral progesterone for the first 12 days of each month.
  Other Names: Evenity
  Arms: Romosozumab
Drug: Placebo — Identical to romosozumab but inactive. This group will also receive a 100-microgram transdermal estradiol patch applied twice weekly, and 200 mg of oral progesterone for the first 12 days of each month.
  Arms: Placebo
Drug: Zoledronic acid — One intravenous infusion
  Other Names: Zoledronate, Reclast
  Arms: Placebo; Romosozumab

SUMMARY:
The goal of this study is to determine whether romosozumab will improve bone density in girls and women with functional hypothalamic amenorrhea (cessation of the menstrual period due to intense exercise, stress, or an eating disorder) who have low bone density. Participants will be randomly assigned to receive romosozumab or placebo for 6 months. All participants will receive one IV infusion of zoledronate at the 6 month visit. All participants will also receive transdermal estradiol and cyclic progesterone. We will investigate whether participants who receive active romosozumab will demonstrate greater improvements in bone density at one year than those who receive placebo. We will also compare bone density over a year with healthy controls (girls and women of similar age who have regular menstrual periods).

ELIGIBILITY:
Inclusion Criteria:

For FHA and controls:

* Female, age 14-30 years, skeletally mature with bone age ≥ 12 years
* For women of reproductive age, agree to use an effective non-hormonal contraceptive method or a progestin releasing intrauterine device (no evidence of systemic skeletal effects) or implant for the study duration
* Biochemical criteria:
* Negative βHCG (pregnancy test)
* TSH within twice the upper limit of normal; potassium, magnesium within the normal range; prolactin <10 ng/mL above the upper limit of normal; FSH not elevated.
* Serum ALT ≤ 3 times upper limit of normal, LDL ≤ 190 mg/dl
* eGFR ≥ 30ml/minute
* If the diagnosis of FHA is unclear, we may check additional labs (e.g., testosterone and sex hormone binding globulin if there is a suspicion of PCOS based on clinical hyperandrogenism).

Additional inclusion criteria for FHA:

* Less than 3 menses in the preceding 6 months
* BMD Z-score ≤ -1.0 at ≥ 1 skeletal site (for subjects <18 years old, we will use the height Z-score-adjusted BMD Z-score using the pediatric bone density calculator developed by the National Institutes of Health and currently maintained by the Children's Hospital of Philadelphia)
* Dental check-up within the past year
* If the menstrual status of the subject is unclear due to the presence of a progestin-releasing IUD, serum estradiol levels will be checked twice, at least one week apart. Both estradiol levels must be < 50 pg/mL.

Exclusion Criteria:

For FHA and controls

* Disease other than FHA known to affect bone, including untreated thyroid dysfunction, Cushing's disease, renal failure, diabetes mellitus
* Use of bisphosphonates
* Use of other medications known to affect bone metabolism within 3 months of the study (other than calcium and vitamin D supplementation).
* Current use of systemic corticosteroids
* Migraine with aura.
* Personal history of or first-degree relative with unprovoked thromboembolism (unless the subject has been tested and ruled out for a hypercoagulable state).
* Active substance use disorder; currently smokes or vapes
* History of malignancy or Paget disease of bone
* Pregnant, planning to become pregnant within 12 months after the end of treatment and/or breastfeeding

Additional exclusion criteria for FHA

* Cardiovascular: History of myocardial infarction or stroke; history of hypertension or use of anti-hypertensive medications
* Immunodeficiency or taking immunosuppressive therapy
* Other conditions that can cause oligo-amenorrhea such as PCOS, primary ovarian insufficiency
* Dental: Osteonecrosis of the jaw (ONJ) or risk factor for ONJ, such as invasive dental procedures (tooth extraction, dental implants, oral surgery in the past 3 months), poor oral hygiene, periodontal and/or pre-existing dental disease
* Planned invasive dental procedure or other planned major surgery for 18 months after the baseline visit
* Known sensitivity or absolute contraindication to any of the products or components of the medications to be administered (romosozumab, zoledronic acid, transdermal estradiol, micronized progesterone, calcium or vitamin D supplements)
* Concerning EKG findings for ischemia

Additional exclusion criteria for normal-weight healthy controls

• BMD Z-score <-2.5 (who we will refer for evaluation)

Ages: 14 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Lumbar spine bone density | 0 and 6 months
  6-month change in lumbar spine bone density
Tibial cortical thickness | 0 and 6 months
  6-month change in tibial cortical thickness
Tibial failure load | 0 and 6 months
  6-month change in tibial failure load

SECONDARY OUTCOMES:
Femoral neck and total hip bone density | 0, 6, and 12 months
  6- and 12-month change in femoral neck and total hip bone density
Lumbar spine bone density | 0 and 12 months
  12-month change in lumbar spine bone density
Radial cortical thickness | 0, 6, and 12 months
  6- and 12-month change in radial cortical thickness
Tibial cortical thickness | 0 and 12 months
  12-month change in tibial cortical thickness
P1NP and CTX | 0, 1, 6, and 12 months
  1-, 6-, and 12-month change in P1NP and CTX
Radial failure load | 0, 6, and 12 months
  6- and 12-month change in radial failure load
Tibial failure load | 0 and 12 months
  12-month change in change in tibial failure load
Lumbar spine, femoral neck, and total hip bone density | 0, 6, and 12 months
  6- and 12-month in lumbar spine, femoral neck, and total hip bone density
P1NP and CTX | 0, 1, 6 and 12 months
  1-, 6- and 12-month change in markers of bone metabolism
Tibial and radial cortical thickness | 0, 6 and 12 months
  6- and 12-month change in tibial and radial cortical thickness
Tibial and radial failure load | 0, 6 and 12 months
  6- and 12-month change in tibial and radial failure load

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Virginia Medical Center, Charlottesville, Virginia